CLINICAL TRIAL: NCT06733428
Title: TRK-3 Agreement and Precision of Pachymetry Function
Brief Title: Agreement and Precision Study
Status: Completed | Type: Observational
Sponsor: Topcon Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: THQ-THINC-2024-01
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Eye Abnormalities; Normal Eyes
MeSH Terms: conditions — Eye Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Normal: Subjects with healthy cornea
  Interventions: Device: Pachymeter
- Cornea: Subjects with abnormal cornea
  Interventions: Device: Pachymeter
- Glaucoma: Subjects with glaucoma
  Interventions: Device: Pachymeter

INTERVENTIONS:
Device: Pachymeter — Measure the thickness of the cornea
  Other Names: TRK-3 auto kerato-refracto tonometer

SUMMARY:
To evaluate the performance of pachymetry function

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary written consent
* Age at least 22 years old
* For glaucoma group only, visual field defect and optic nerve damage consistent with glaucoma
* For cornea group only, cornea abnormality

Exclusion Criteria:

* Ocular condition that may affect ability to perform cornea measurements
* Have or is suspected to have ocular infection
* Unable to tolerate eye testing

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects seeing an eye doctor that have normal cornea, cornea abnormality, or glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Cornea thickness | 1 day
  thickness of the cornea

CONTACTS AND LOCATIONS:
Locations (1):
- Illinois College of Optometry, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No